CLINICAL TRIAL: NCT01428076
Title: An Open-Label Single-Center Study in Patients With Great Saphenous Vein Incompetence to Investigate the Pharmacokinetic Properties of Polidocanol Endovenous Microfoam (PEM)
Brief Title: Pharmacokinetic Study of Polidocanol Endovenous Microfoam (PEM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAP.VV008
Record Dates: First submitted 2011-08-30; First posted 2011-09-02 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Varicose Veins
Keywords: Varicose Veins; SFJ Reflux
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose Polidocanol Endovenous Microfoam (Experimental)
  Interventions: Drug: Polidocanol Endovenous Microfoam (PEM)
- Medium Dose Polidocanol Endovenous Microfoam (Experimental)
  Interventions: Drug: Polidocanol Endovenous Microfoam (PEM)

INTERVENTIONS:
Drug: Polidocanol Endovenous Microfoam (PEM) — Pharmacokinetic comparison of different doses of drug

SUMMARY:
Varicose veins are enlarged, noticeably bulging veins, which commonly occur in the legs and may cause discomfort. In this study, patients with varicose veins in the legs will be participating. The purpose of this research study is to evaluate the pharmacokinetic profile of two different doses of an investigational drug, Polidocanol Endovenous Microfoam (PEM), an investigational treatment for varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; age 18 to 75 years
* Superficial venous disease where SFJ incompetence is the predominant source of reflux (reflux > 0.5 seconds on duplex ultrasonography) associated with incompetence of the great saphenous vein (GSV) or other major accessory vein
* Expected need for microfoam of 10 mL to fill the incompetent GSV and tributaries (minimum trunk vein diameter of 6mm)
* Clinically normal renal and hepatic function on serum chemistry
* Ability to comprehend and sign an informed consent document in English

Exclusion Criteria:

* Major co-existing disease (e.g. malignancy; pulmonary disease; renal or hepatic insufficiency; serious skin disease/condition that may compromise the ability of the patient to comply with the compression protocol, etc.)
* Clinically significant abnormal ECG or clinical condition which may affect interpretation of ECG, for example, history of Long QT Syndrome, Brugada Syndrome, electronic cardiac pacemaker, chronic atrial fibrillation, recent myocardial infarction or congestive heart failure.
* Patients taking QT prolonging medications
* Any of the following findings on screening ECG:
* QRS > 110 ms
* HR < 45 bpm
* HR > 100 bpm
* QTcF > 470 ms
* PR > 220 ms
* Patients who only have telangiectatic or reticular veins (Clinical Finding C1, as assessed by CEAP Classification of Venous Disorders)
* Leg obesity impairing the ability to access the vein to be treated and/or to apply post-procedure compression bandaging and stockings
* Ultrasonographic or other evidence of current or previous deep vein thrombosis or occlusion
* Deep venous reflux unless clinically insignificant in comparison to superficial reflux
* Peripheral arterial disease precluding the wearing of post-procedure compression bandaging and stockings
* Reduced mobility (unable to walk unaided for 5 minutes per waking hour)
* History of deep vein thrombosis, pulmonary embolism or stroke, including evidence of prior DVT on duplex ultrasound
* Major surgery, prolonged hospitalization or pregnancy within 3 months of screening
* Known allergic response to polidocanol or heparin, including history of heparin-induced thrombocytopenia, and/or multiple allergic reactions
* Current alcohol or drug abuse
* Pregnant or lactating women
* Women of childbearing potential not using effective contraception for at least one month prior to study enrollment (i.e., treatment) and/or unwilling to continue birth control until Visit 4
* Participation in a clinical study involving an investigational pharmaceutical product or device within the 3 months prior to screening
* Previous treatment with Polidocanol Endovenous Microfoam (PEM) in a previous PEM study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular and Vein Center of Florida, Bradenton, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Polidocanol 1%: polidocanol injectable foam 1% concentration
- Polidocanol 2%: polidocanol injectable foam 2% concentration
Period: Overall Study
Arm/Group | Polidocanol 1% | Polidocanol 2%
Started | 9 | 12
Completed | 9 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Polidocanol 2%: polidocanol intravenous foam 2% concentration
- Total: Total of all reporting groups
Arm/Group | Polidocanol 1% | Polidocanol 2% | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (9.62) | 49.9 (11.4) | 51.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (2.52) | 27.1 (5.19) | 27.1 (4.16)

OUTCOME MEASURES:

1. Primary Outcome: Weight-adjusted Polidocanol Cmax (Serum)
Description: Cmax measured and adjusted for weight
Time Frame: pharmacokinetics measured- predose, 1, 4, 5, 7, 9, 11, 14, 15, 17, 20, 25, 30 minutes post dose, 1, 2, 3, 4, 5, 6, 8 hours post dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Males-polidocanol 1%; Females-polidocanol 1%: polidocanol injectable foam 1% concentration
- Males-polidocanol 2%; Females- Polidocanol 2%: polidocanol injectable foam 2% concentration
Arm/Group | Males-polidocanol 1% | Males-polidocanol 2% | Females-polidocanol 1% | Females- Polidocanol 2%
Number analyzed (Participants) | 3 | 6 | 6 | 5
ng/mL | 584.1 (142.8) | 1188.7 (341.7) | 840.7 (437.6) | 1189.6 (331.2)

ADVERSE EVENTS:
Arm/Group | Polidocanol 1% | Polidocanol 2%
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 4/9 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polidocanol 1% (N=9) | Polidocanol 2% (N=12)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Extravasation (General disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 3 (3)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
thrombosis (Vascular disorders) | 0 (0) | 1 (1)
venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No